CLINICAL TRIAL: NCT05943899
Title: Sodium-Glucose co Transporter 2 Inhibitors in Patients With Type 2 Diabetes Mellitus and Moderate to Severe Liver Fibrosis: A Preliminary Retrospective Study
Brief Title: Effect of SGLT-2 Inhibitors in Patients With T2DM and Moderate to Severe Liver Fibrosis
Status: Completed | Type: Observational
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Other Study IDs: CLD&SGLT2
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Type2diabetes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study will be of 12 months duration where 40 T2DM patients coming to FORTIS C-DOC hospital in OPD with F3 fibrosis will be included in the study. The population will be representative of different socio-economic strata of the society. Clinical and dietary profiles, phenotypic markers (acanthosis nigricans, buffalo hump, skin tags, xanthelasma, double chin, arcus, hirsutism) anthropometric assessments body mass index; biochemical markers like liver function test, HbA1c, prothrombin time/INR, and fibroscan will be assessed.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most prevalent cause of chronic liver disease worldwide. Type 2 diabetes mellitus (T2DM) and nonalcoholic fatty liver disease (NAFLD) commonly exist together. The presentations of NAFLD range from simple steatosis (NAFL), nonalcoholic steatohepatitis (NASH), and cirrhosis. NAFLD has a prevalence of 70% among T2DM patients. This results in adverse outcomes such as higher rates of mortality due to cirrhosis. Cirrhosis and liver failure occurs in 11%-20% in NASH patients. Overweight/obesity and insulin resistance (IR) have been strongly linked with NAFLD. Patients with diabetes or prediabetes had progressive fibrosis when their serial biopsies were studied. Those patients with worsening metabolic risk factors tend to have increased progression from NAFL to NASH and fibrosis.

Non-invasive assessment of disease are based on clinical parameters such as age, sex, liver function test, platelet count, lipid profile, body mass index (BMI), and imaging modalities such as ultrasound (USG), transient Elastography (TE), and magnetic resonance imaging (MRI) mass spectroscopy. Fibrosis stage is recognized as the most objective indicator of liver damage and is the best prognostic marker for morbidity and mortality in liver disease of various etiologies. The rise in the incidence of nonalcoholic steatohepatitis (NASH) has necessitated the development of an effective prevention methodology.

Sodium-glucose cotransporter type-2 (SGLT2) inhibitors are glucose-lowering agents that improve glucose control while promoting weight loss and lowering serum uric acid levels. These agents may exert cardiovascular and renal protection in T2DM patients with established cardiovascular disease. Recent findings from both randomized controlled trials and open-label studies have also shown that SGLT2 inhibitors are able to reduce fatty liver content, as assessed by different imaging techniques, and improve biological markers of NAFLD, especially serum liver enzymes, in patients with T2DM. In addition, there are emerging data to suggest a mechanism beyond the reduction of hyperglycaemia and body weight, and a potential role for the decrease in low-grade inflammation and oxidative stress associated with SGLT2 inhibitor therapy. This positive effect of SGLT2 inhibitors on NAFLD complements their already well-known effects on cardiovascular and chronic kidney diseases.

SGLT2 inhibitors significantly reduced liver fat when added to the standard treatment for T2DM. There are very few studies which have examined the effects of SGLT2 inhibitors in patients with F3 fibrosis. In a randomized controlled trail addition of 5mg/d dapagliflozin(SGLT2 inhibitor) for 24 weeks decreased liver stiffness measure from 14.7 to 11 kPa and also reduced visceral fat. In a prospective non-randomized study 100mg canagliflozin (SGLT-2 inhibitor) administered once daily for 12 months significantly reduced hepatic fat 17.6 to 12 after 6 months measured by magnetic resonance imaging. It also reduced body fat and improved liver enzymes. Another study showed reduction in patients with F4 fibrosis with exenatide once weekly and dapagliflozin once daily at 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients with T2DM having F3 fibrosis/Child's A Cirrhosis

Exclusion Criteria:

1. Type 1 Diabetes
2. Alcohol consumption per day (Men >20 g and women >10 g)
3. Patients with Child B or Child C Cirrhosis
4. Known case of HIV infection
5. Congestive heart disease
6. Positive hepatitis B or hepatitis C, secondary causes of fatty liver (eg, consumption of amiodarone and tamoxifen) and congestive hepatopathy.
7. Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM patients visiting Fortis CDOC hospital and diagnosed with Moderate/Severe fibrosis were included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Association between SGLT2i intake and hepatic fibrosis | 12 months
  T2DM patient with moderate to severe fibrosis given SGLT2i and then again evaluated during follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Fortis CDOC Hospital
Locations (1):
- Fortis CDOC Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No